CLINICAL TRIAL: NCT06363006
Title: Evaluation of the Efficacy and Safety of Cardonilimab Injection Combined With TKI as Second-line Treatment for Advanced Hepatocellular Carcinoma: A Single-arm, Open-label, Multicenter Real-world Clinical Study
Brief Title: Combination of Cardonizumab Injection and TKI Second Line Therapy for Advanced Hepatocellular Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23C3280
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TKI+Cardonilizumab (Experimental): TKI:Tyrosine kinase inhibitors can serve as competitive inhibitors of adenosine triphosphate (ATP) binding to tyrosine kinase, as well as analogues of tyrosine, blocking the activity of tyrosine kinase and inhibiting cell proliferation.
  Cardonilizumab:It can block the interaction between PD-1, CTLA-4 and their ligands PD-L1/PD-L2, B7.1/B7.2, thereby blocking the immunosuppressive response of the PD-1 and CTLA-4 signaling pathways, promoting tumor specific T cell immune activation, and inhibiting tumor cell growth.
  Interventions: Drug: TKI+Cardunilimab

INTERVENTIONS:
Drug: TKI+Cardunilimab — Cardonilizumab 6mg/kg, IV, Q2W + lenvatinib 8mg (body weight < 60kg) or 12mg(body weight ≥60kg) PO, QD, / Sorafenib 400mg, PO, BID/ Regorafenib 160mg, PO, QD/ Donafenib 200mg, PO, BID。 omniscience

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of cardonilizumab injection combined with TKI in second-line treatment of advanced hepatocellular carcinoma. The main questions it aims to answer are:

* Objective response rate (ORR) for evaluation
* Disease Control Rate (DCR); Duration of relief (DoR); Progression free survival (PFS); Total survival time (OS); Safety。

DETAILED DESCRIPTION:
Have received at least one prior systemic treatment progression or intolerance for HCC. Cardonilizumab was administered every 2 weeks on the first day of each cycle for up to 24 months in the absence of investigator judgment that there is no longer a clinical continuation benefit, intolerable toxicity, initiation of a new antitumor therapy, withdrawal of informed consent, loss of follow-up, death, or other protocol requirements for treatment termination. Cardonilizumab will complete infusion within 60 minutes (± 10 minutes). Continuous monitoring of potential infusion reactions and allowing pre-treatment of hypersensitivity reactions or infusion rate adjustment according to protocol guidelines. For subjects who cannot tolerate a 60-minute infusion, the infusion time can be extended up to 120 minutes. Dose adjustment of cardonilizumab is not allowed during treatment, but delayed dosing is allowed for up to 12 weeks (since the last dosing time). If glucocorticoids are used in the treatment of irAE, In both cases where the glucocorticoid reduction process resulted in the suspension of cardonilizumab for more than 12 weeks, or in the treatment of AE that may or may not be related to cardonilizumab, and where the investigator determined that the patient would benefit from continued treatment, permission to continue treatment was required after discussion with the sponsor medical Ombudsman.

ELIGIBILITY:
Inclusion Criteria:Participants must meet all of the following inclusion criteria to be admitted to the study:

1. Patients with histologically/cytologically confirmed hepatocellular carcinoma or cirrhosis meet the clinical diagnostic criteria of the American Association for the Study of Liver Diseases (AASLD) for hepatocellular carcinoma.
2. Age ≥18 and ≤75 years old.
3. ECOG physical status score 0 or 1.
4. Barcelona Clinic Liver Cancer (BCLC) stage C; It is not suitable for radical surgery and/or local treatment or stage B that progresses irremediably after surgery and/or local treatment.
5. Progression or intolerance after receiving at least one systemic antitumor therapy for hepatocellular carcinoma prior to initial administration
6. According to RECIST v1.1, there is at least one untreated measurable lesion or one that has been locally treated (e.g., Measurable lesions with clear progression (RECIST v1.1 standard) after radiofrequency ablation, injection of anhydrous ethanol or acetic acid, cryoablation, high-intensity focused ultrasound, transarterial embolization chemotherapy, transarterial embolization, etc., can be measured repeatedly.
7. Child-Pugh Level A.
8. Any treatment-related toxicity (due to prior treatment) must be resolved to baseline or stable prior to enrollment, except for hair loss.

Exclusion Criteria:Participants who meet any of the following criteria will not be eligible to participate in the study:

1. Fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma and other components previously confirmed by histology/cytology.
2. History of hepatic encephalopathy.
3. History of liver transplantation.
4. There is clinically significant pericardial effusion; There are clinical symptoms of a pleural effusion requiring drainage.
5. Clinically significant ascites are defined as meeting the following criteria: ascites can be detected by physical examination during screening or ascites need to be drained during screening.
6. Co-infection with HBV and HCV (a history of HCV infection but negative HCV RNA can be considered not infected with HCV).
7. There is central nervous system metastasis or meningeal metastasis.
8. Bleeding from esophageal or fundus varices caused by portal hypertension occurred within 6 months before the first dose Event. A gastroscopy must have been performed within 6 months prior to initial dosing, and participants with severe (G3) varicose veins were not allowed to participate in the study.
9. Patients with any physical signs or history of bleeding, regardless of severity; Patients with any bleeding or bleeding event ≥CTCAE grade 3 within 4 weeks prior to initial dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR Full single-arm, open, multicenter prospective clinical study | 3 years
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.
Progression-free Survival (PFS) | 1.5 years
  A duration from the date of initial treatment with TKI plus Cardonizumab to disease progression (defined by RECIST 1.1) or death of any cause.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 3 years
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Overall Survival (OS) | 3 years
  Duration from the date of initial treatment with TKI plus Cardonizumab to the date of death due to any cause.
Duration of Response (DOR) | 3 years
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Stable Disease (SD) | 3 years
  Proportion of patients with stable disease status more than 4 months.
Progression free survival rate | 1.5 years
  Portion of patients who do not experience disease progression (defined by RECIST 1.1) or death of any cause after treated with TKI plus Cardonizumab for 3 months and 6 months, respectively.

OTHER OUTCOMES:
Any adverse events related with treatment with TKI plus Cardonizumab. | 3 years
  Safety and tolerability of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital (CAMS&PUMCH), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No